CLINICAL TRIAL: NCT04815421
Title: Therapeutic Efficacy of Dredging Three Yang Meridians of Hand With Deep Tissue Massage on Stiff-neck Syndrome
Brief Title: Deep Tissue Massage on Stiff-neck Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zhanglingyun
Record Dates: First submitted 2021-03-09; First posted 2021-03-25 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Massage; Meridian; Pain
Keywords: meridian; massage; stiff-neck syndrome; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Patients who were diagnosed with stiff-neck syndrome according to the diagnostic criteria（Acute onset of severe pain and stiffness in one-sided neck after sleep; Mostly because of bad sleep posture or cold in neck, shoulder or head; Pain or discomfort can radiate to head, arm and back; Any attempt to move neck can obviously exacerbate the pain; The head slants to the affected side; Without neck injury history or other relative systematic diseases.; Neck X-ray film has no positive signs such as degenerative lesions of cervical spine; Trachelismus and rhomboideus major/ minor, levator scapulae accessible lumps or streak in muscle. All criteria conformed to the prescription in criteria of diagnostic and therapeutic effect of orthopaedic and traumatologic diseases and syndromes in traditional Chinese medicine）. They were randomly enrolled in meridian group or paste group according to the visiting time (with digital random table).
Who Masked: Outcomes Assessor
Masking Description: Two persons of our protocol who was unknown of the patients' treatment method and period estimated the VAS of every patient freely and evaluated the clinical effects and outcomes according to the criteria of diagnostic and therapeutic effect of orthopaedic and traumatologic diseases and syndromes in traditional Chinese medicine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the paste group (Experimental): Patients in the paste group were treated with Nanxing paste on the affected region include shoulder, neck or back and no more than 3 pieces. The therapy duration was 6 days.
  Interventions: Other: the paste group
- the meridian group (Experimental): Patients in the meridian group were treated with dredging the same side Hand yang meridian techniques
  Interventions: Other: the meridian group

INTERVENTIONS:
Other: the paste group — Patients in the paste group were treated with Nanxing paste on the affected region include shoulder, neck or back and no more than 3 pieces. The paste lasted for 24 hours and then peeled it rested the pasted region for 24 hours and changed another paste on the pain region. The therapy duration was 6 days.
  Arms: the paste group
Other: the meridian group — Patients in the meridian group were treated with dredging the same side three yang meridian techniques(include the gliding techniques of deep tissue massage on three yang meridians of back hand (the second, fourth and fifth metacarpal bone); pinching and kneading the second, fourth and fifth phalanges of fingers of the affected side hand; Encourage the patient to try his best to roll his neck to the most tolerable degree during dredging the meridian) and the total time was about 3 to 5 minutes according the tolerance of every patient . The massage will not stop until the meridian route was relatively smooth, soft and thermal or light red. The sequence of massage is Hand Yangming meridian(LI) the first, Hand Taiyang meridian(SI) the second and Hand Sanjiao(SJ) the last. The frequency of massage was once a day.
  Arms: the meridian group

SUMMARY:
This is a randomized controlled study . The objective is to observe the therapeutic effects of dredging three yang meridians of hand with deep tissue massage on stiff-neck syndrome.

Methods: patients with stiff-neck syndrome were randomly divided into meridian group and paste group.The meridian group were treated once a day for 3 days and the paste group therapy was a 3 courses therapy（ one course includes 24-hour rest and 24-hour paste）. After 3 courses, pain was assessed by visual analogue scale (VAS), the therapeutic effects were compared between the two groups in every stage of the therapy and the self-controlled study.The evaluation criteria on stiff-neck syndrome is based on criteria of diagnostic and therapeutic effect of orthopaedic and traumatologic diseases and syndromes in traditional Chinese medicine . Cure: Absence of neck-stiff, neck sore and free functional activities. Improvement: partially functional activities with light to moderate pain. Failure: No improvement or alleviation of neck stiff and agony. All data will be analyzed by SPSS 16.0, the statistical difference is considered if the P<0.05 and the significant difference is considered if the P<0.01 .

DETAILED DESCRIPTION:
1 Clinical Materials 1.1 Diagnostic criteria Acute onset of severe pain and stiffness in one-sided neck after sleep; Mostly because of bad sleep posture or cold in neck, shoulder or head; Pain or discomfort can radiate to head, arm and back; Any attempt to move neck can obviously exacerbate the pain; The head slants to the affected side; Without neck injury history or other relative systematic diseases.; Neck X-ray film has no positive signs such as degenerative lesions of cervical spine; Trachelismus and rhomboideus major/ minor, levator scapulae accessible lumps or streak in muscle. All criteria conformed to the prescription in criteria of diagnostic and therapeutic effect of orthopaedic and traumatologic diseases and syndromes in traditional Chinese medicine.

1.2 Inclusion criteria The onset of symptoms and signs are less than 24 hours; Male or female aged from 14 to 60 years; No other therapy before grouped; Be willing to participate the study and sign the informed consent.

1.3 Exclusion criteria Stiff neck patients who had diagnosed cervical vertebra or cervical spondylosis; Suffered from systemic collagen immune diseases or other acute or chronic infection; Use pain-killer drugs may affect the outcome evaluation; Refuse to join the trial; Drop out in follow-up visit; Aggravation of disease or complications during the study.

1.4 Patients All patients were outpatients and be diagnosed with stiff-neck syndrome according to the diagnostic criteria. They were randomly allocated into 2 groups (meridian group and paste group) according to the visiting time (with digital random table)and their wills.

2.1 meridian group Patients in the meridian group were treated with dredging the same side three yang meridians of hand techniques(include the gliding techniques of deep tissue massage on the three yang meridians of back hand (the second, fourth and fifth metacarpal bone); pinching and kneading the second, fourth and fifth phalanges of fingers of the affected side hand; Encourage the patient to try his best to roll his neck to the most tolerable degree during dredging the meridians) and the total time was about 3 to 5 minutes according the tolerance of every patient and the smooth of three yang meridians of hand. The massage will not stop until the meridian route was relatively smooth, soft and thermal. The sequence of massage is Hand Yangming meridian(LI) the first, Hand Taiyang meridian(SI) the second and Hand Sanjiao(SJ) the last. The frequency of massage was once a day.

2.2 paste group Patients in the paste group were treated with Nanxing paste on the affected region include shoulder, neck or back and no more than 3 pieces. The paste lasted for 24 hours and then peeled it rested the pasted region for 24 hours and changed another paste on the pain region. The therapy duration was 6 days.

Pain was assessed by visual analogue scale (VAS), the therapeutic effects were compared between the two groups in every stage of the therapy and the self-controlled study.The evaluation criteria on stiff-neck syndrome is based on criteria of diagnostic and therapeutic effect of orthopaedic and traumatologic diseases and syndromes in traditional Chinese medicine . Cure: Absence of neck-stiff, neck sore and free functional activities. Improvement: partially functional activities with light to moderate pain. Failure: No improvement or alleviation of neck stiff and agony. All data will be analyzed by SPSS 16.0, the statistical difference is considered if the P<0.05 and the significant difference is considered if the P<0.01 .

ELIGIBILITY:
Inclusion Criteria:

* The onset of symptoms and signs are less than 24 hours
* Male or female aged from 14 to 60 years
* No other therapy before grouped
* Be willing to participate the study and sign the informed consent

Exclusion Criteria:

* Stiff neck patients who had diagnosed cervical vertebra or cervical spondylosis
* Suffered from systemic collagen immune diseases or other acute or chronic infection
* Use pain-killer drugs may affect the outcome evaluation
* Refuse to join the trial; Drop out in follow-up visit
* Aggravation of disease or complications during the study

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
clinical effects | day1 to day 6
  cure or improvement or failure(Cure: Absence of neck-stiff, neck sore and free functional activities. Improvement: partially functional activities with light to moderate pain. Failure: No improvement or alleviation of neck stiff and agony)
VAS evaluation between the 2 groups | day1 to day 6
  We used the visual analogue scale(VAS) to evaluate the score of pain score(0=none,10=maximum )

CONTACTS AND LOCATIONS:
Overall Officials: Lingyun Zhang, Master, Study Chair — The Affiliated Hospital of Qingdao University; Xue Jing, Doctor, Principal Investigator — The Affiliated Hospital of Qingdao University; Xiaoju Peng, Doctor, Principal Investigator — The Affiliated Hospital of Qingdao University; Ying Liu, no, Study Director — The Affiliated Hospital of Qingdao University; Xueguo Sun, Doctor, Study Director — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No